CLINICAL TRIAL: NCT04153331
Title: Burden of Influenza at Emergency Department Level : BIED
Acronym: BIED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0755
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2020-01

CONDITIONS: Emergencies; Flu
MeSH Terms: conditions — Emergencies; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients admitted to emergency department with medical cause (Experimental): Patient included in emergency with a nasal swab
  Interventions: Other: Nasal swab

INTERVENTIONS:
Other: Nasal swab — Patient included in emergency with a nasal swab

SUMMARY:
Seasonal influenza surveillance in France relies on several sources to detect the onset of the epidemic early, as well as to estimate the severity of epidemics and their impact on the health system. However, the data collected do not fully measure the impact of epidemics on the hospital system.

Increasing the investigator's knowledge of the impact of influenza on the hospital system, particularly on emergencies, which are the most affected service, is essential to better adapt the resources put in place to care for patients.

The study will allow a better understanding of the influenza burden, by systematically documenting the severe events (i.e. requiring consultations to the Emergency Rooms) that are triggered by influenza but not necessarily reported/recorded as influenza.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Consultation for a medical cause

Exclusion Criteria:

* Consultation for a non-medical cause (trauma...)
* Pregnant, parturient and lactating women
* Persons deprived of their liberty
* Persons of full age who are subject to a legal protection measure
* Persons not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2487 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Proportion of laboratory confirmed influenza among patients admitted to Emergency Room during the influenza season | 1 day (at admission)
  The proportion of laboratory confirmed influenza cases will be calculated by dividing the number of patients with laboratory confirmed influenza by the total number of patients included

SECONDARY OUTCOMES:
Proportion of patients with co-morbidities | 1 day (at admission)
  to evaluate the proportion of patients consulting emergency department who have co-morbidities according to the result of the virological sampling
Proportion of patients with laboratory confirmed influenza and related outcomes | 1 day (at admission)
  to estimate the proportion of patients with a laboratory confirmed influenza stratified on the emergency department visit outcomes (hospitalization in medicine, hospitalization in intensive care unit or return home) and other covariates
Proportion of patients who consult for other causes than influenza | 1 day (at admission)
  to estimate the proportion of patients with a laboratory confirmed influenza consulting for other causes than influenza
Proportion of asymptomatic influenza cases among patients with laboratory confirmed influenza | 1 day (at admission)
  The proportion asymptomatic influenza cases will be calculated by dividing the number of patients with asymptomatic influenza by the total number of laboratory confirmed influenza

CONTACTS AND LOCATIONS:
Overall Officials: Philppe VANHEMS, MD, Principal Investigator — Service Hygiène, Epidémiologie et Prévention
Locations (1):
- Service Hygiène, Epidémiologie et Prévention, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amour S, Rubio AP, Orsi A, Oppert M, Loebermann M, Del Pozo Vegas C, Tazarourte K, Douplat M, Jacquin L, Icardi G, Walker J, Glass A, Nealon J, Chaves SS; FERS Study Group; Bricout H, Vanhems P. Influenza in Adults Seeking Care at Seven European Emergency Departments: A Prospective Active Surveillance During the 2019-2020 Influenza Season. Influenza Other Respir Viruses. 2024 Nov;18(11):e70040. doi: 10.1111/irv.70040. PMID 39568106